CLINICAL TRIAL: NCT05961930
Title: Surgeon's Performance in Predicting Postoperative Infections
Acronym: SPIRIT
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Sesmu M. Arbous, MD PhD MSc, Principal Investigator, Sesmu M. Arbous, MD PhD MSc, Leiden University Medical Center
Other Study IDs: 2022-64
Record Dates: First submitted 2023-03-03; First posted 2023-07-27 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Infection
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Surgeons estimate of postoperative infection: All surgeons will be asked to fill in a questionnaire, containing 5 questions, pertaining to the estimated risk of postoperative infection (within 30days). Thus there is a single arm and no comparison.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Surgeons will be asked to fill in a short questionnaire after surgery on risk of postoperative infection

SUMMARY:
Post-surgical (bacterial) infections are the most frequent post-surgical complications, including deep or superficial wound infections, urinary tract infections, pneumonia, and even sepsis. Approximately 6.5-25% of all surgical patients will develop any type of bacterial infection. To personalize surgical infection management, (Artificial Intelligence) models are in the making to predict which patients are at high or low risk of developing a post-surgical infection. In order to benchmark these prediction models to the predictive capabilities of surgeons, the investigators aim to investigate the performance of surgeons in predicting the risk of a patient developing (any type) of post-surgical infection within 30 days.

DETAILED DESCRIPTION:
A prospective non-interventional study is performed to collect surgeons' predictions on the risk of a patient developing a postoperative infection within 30 days of surgery. Surgeons are asked to fill in a short questionnaire asking about the estimated infection risk. The actual outcome (infection < 30 days of surgery) of a patient will be collected retrospectively after completion of the study. This study will have no effect on standard care: surgical interventions and postoperative care will be carried out according to standard clinical practice. Besides a one-time estimate of the surgeon, immediately after the surgical procedure, no other interventions will be performed and surgical specialists will carry out their normal post-surgical care, including screening and treating (if necessary) their patients for postoperative infections.

ELIGIBILITY:
Predictions are made for patients with the following inclusion and exclusion criteria:

Inclusion Criteria:

* Adult patients (>18 years old)
* Acute or elective surgery
* Invasive or minimally invasive surgical procedures

Exclusion Criteria:

* Outpatient procedures or procedures not requiring any form of monitoring/anesthesia
* Procedures for which the primary indication is (treatment for) an infection
* Radiological procedures
* Cardiological catheterization procedures
* Psychiatric treatment under anaesthesia (i.e. electroconvulsive therapy)
* Sole anaesthetic procedures except for implantation of a neurostimulator
* Brachytherapy procedures
* Endoscopic procedures for diagnostic purposes only
* Procedures that only entail the taking of a biopsy for diagnostic purposes
* Patients that are pregnant
* Procedures out of office hours (before 8.00 am or after 5.00 pm)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, surgical population of different surgical subspecialties.
Sampling Method: Non-Probability Sample
Enrollment: 594 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
The discriminative predictive performance of surgeons with respect to estimating the risk of developing (any type) bacterial post-surgical within 30 days of surgery | 30 days
  The primary outcome measure of discrimination are area under the receiving operating characteristic curve (AUROC). Predictions are compared to the occurrence of a postoperative infection requiring treatment, surgical intervention or registration within 30 days of surgery.
The calibration properties of surgeons with respect to estimating the risk of developing (any type) bacterial post-surgical within 30 days of surgery | 30 days
  Calibration plots with slope and intercept

SECONDARY OUTCOMES:
Relationship between the certainty in estimate and the predictive performance of surgeons | 30 days
  Surgeons are questioned on their certainty in the provided estimate
Relationship between patient factors and predicted risk | 30 days
  Surgeons are questioned to indicate for a list of patient factors whether they were of impact to the decision
Predictive performance per surgeons and patients subgroups | 30 days
  Surgeons subgroups are based on specialty, years of experience, level of experience, sex. Patient subgroups include, surgical specialty, age groups, type of surgical procedure, planned or emergency intervention.
Relationship between predicted risk of surgeons and if they perform additional actions | 30 days
  Surgeons are asked to indicate whether they performed additional actions for this patient in the questionnaire.
Comparison between the predicted risk of surgeons and an artificial intelligence algorithm | 30 days
  The performance of the physicians is compared to that of the artificial intelligence algorithm by means of AUROC

CONTACTS AND LOCATIONS:
Locations (1):
- Sesmu Arbous, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No